CLINICAL TRIAL: NCT03213353
Title: A SingleDose Rand, TwoPeriod, Crossover Bioequivalence Study Between a Combination Tablet With Paracetamol, Guaifenesin and Penylephrine HCL (Wrafton Lab Ltd, UK) and Vicks Active SymptoMax Plus, Powder for Oral Solution (Wrafton Lab Ltd, UK) in Healthy Adult Volunteers
Brief Title: A Bioequivalence Study Between Two Brands of Medications to Treat Cough & Cold Symptoms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CO-160408130708-URCT
Record Dates: First submitted 2017-06-20; First posted 2017-07-11 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Bioequivalence; Healthy Volunteers
MeSH Terms: interventions — Guaifenesin; Oxymetazoline; Powders; Solutions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment sequence AB (Experimental): Treatment A (experimental): Two tablets of Combination tablet with paracetamol, guaifenesin and phenylephrine hydrochloride each containing 250 mg paracetamol, 100 mg guaifenesin, and 5 mg phenylephrine hydrochloride
  Treatment B (active comparator): One sachet Vicks Active SymptoMax Plus, powder for oral solution, containing 500 mg paracetamol, 200 mg guaifenesin, and 10 mg phenylephrine hydrochloride
  Interventions: Drug: Tablet paracetamol, guaifenesin and phenylephrine HCL; Drug: Vicks Active SymptoMax Plus powder for oral solution
- Treatment sequence BA (Experimental): Treatment A (experimental): Two tablets of Combination tablet with paracetamol, guaifenesin and phenylephrine hydrochloride each containing 250 mg paracetamol, 100 mg guaifenesin, and 5 mg phenylephrine hydrochloride
  Treatment B (active comparator): One sachet Vicks Active SymptoMax Plus, powder for oral solution, containing 500 mg paracetamol, 200 mg guaifenesin, and 10 mg phenylephrine hydrochloride
  Interventions: Drug: Tablet paracetamol, guaifenesin and phenylephrine HCL; Drug: Vicks Active SymptoMax Plus powder for oral solution

INTERVENTIONS:
Drug: Tablet paracetamol, guaifenesin and phenylephrine HCL — Each subject will receive two tablets, each containing 250 mg paracetamol, 100 mg guaifenesin, and 5 mg phenylephrine hydrochloride
  Other Names: Benylin Cough & Cold All in One Relief Tablets
Drug: Vicks Active SymptoMax Plus powder for oral solution — Each subject will receive one sachet, containing 500 mg paracetamol, 200 mg guaifenesin, and 10 mg phenylephrine hydrochloride

SUMMARY:
This is a single-dose, randomized, two-period cross-over study with 72 healthy male and female volunteers. The investigational products will be given (after fasting overnight) at separate visits separated by 7 ± 3 days. Blood for pharmacokinetic analyses will be drawn pre-dose and at 5, 10, 15, 20, 25, 30, 40, 60, 75, 90, 105 minutes, as well as 2, 2.25, 3, 4, 5, 6, 8, and 12 hours after drug administration. Subjects will also be monitored to capture any adverse events that may occur. Bioequivalence will be assessed based on the single-dose pharmacokinetics of paracetamol, guaifenesin and phenylephrine, respectively

ELIGIBILITY:
Inclusion Criteria:

1. Subjects being verified as "Healthy": "Healthy" is defined as absence of any diseases or abnormalities on the basis of physical examination, standard clinical laboratory, and instrumental examinations performed at the screening visit.
2. Females of childbearing potential must have a negative urine pregnancy test at the baseline visit.
3. Male or non-pregnant, non-lactating female agree to the contraceptive requirements (including female partner's use of a highly effective method of birth control for at least 3 months before the study, during the study, and for 30 days after the last dose of study drug) as outlined in Section 11.6 (Note: Female subjects are not permitted to use hormonal contraceptives as per exclusion criterion 7).
4. Body Mass Index (BMI) between 18.5 and 30.0 kg/m2, inclusive, and a total body weight of at least 50.0 kg.
5. Volunteers who agree to abstain from alcohol consumption for at least 48 hours prior to dosing and until the last blood sample collection of each study period.

Exclusion Criteria:

1. Use of medications, including prescription medication, over-the-counter medication including vitamins, herbal supplements, medicinal plants (e.g., supplements containing garlic extract), and topical preparations of drugs that are systemically absorbed (e.g., steroids and non-steroid anti-inflammatory drugs) within two weeks prior to dosing.
2. Use of St. John's wort (Hypericum perforatum) within 30 days prior to dosing.
3. Depot injection or an implant of any drug within 3 months prior to dosing.
4. Abnormal results of laboratory and instrumental methods of examinations, including electrocardiogram (ECG).
5. Is hypersensitive, intolerant, or has experienced an allergic reaction to the active ingredients or excipients of drug products that will be used for the study, or has had severe allergy (e.g., anaphylaxis, angioedema) in the past.
6. Females with a positive pregnancy test and/or are breast-feeding.
7. Females, currently using hormonal contraceptives (including use less than 2 months prior to enrollment).
8. Males with a pregnant spouse or partner or males who are not willing to prevent conception in a spouse or partner.
9. History of regular alcohol consumption in the 6 months before screening, exceeding weekly limits of 10 alcohol units (2 L of wine or 5 L of beer or 0.5 L of spirits) or presence of information on alcoholism, substance, or drug abuse in medical history.
10. Alcohol consumption within 48 hours prior to dosing, positive respiratory alcohol test at screening, or inability to abstain from alcohol consumption until the last blood sample collection of each study period.
11. Volunteers who smoke more than 10 cigarettes per day or have an uncontrollable habit of chewing or inhaling nicotine products.
12. Drug addiction in history, or a positive urine test for psychoactive or narcotic substances.
13. Use of caffeine products exceeding 500 mg caffeine daily (5 cups of coffee) and the inability to abstain from caffeine products within 48 hours before dosing and prior to the last blood sample collection of each study period.
14. Use of xanthine containing products (e.g., coffee, tea, chocolate, or cola drink) within 48 hours before dosing and prior to the last blood sample collection of each study period.
15. Ingestion of food or beverages containing grapefruit, Chinese grapefruit (pomelo), or Seville oranges (including marmalade) within 10 days prior to the first dose of the investigational product and inability to stop taking these products during the study.
16. Positive test for human immunodeficiency virus (HIV) 1 or 2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (anti-HCV) or syphilis (RW).
17. Heart rate <60 or >90 per minute at rest, or systolic blood pressure <100 or >130 mm Hg, or diastolic blood pressure <70 or >90 mm Hg.
18. Clinically significant signs and symptoms or history of respiratory, cardiovascular, gastrointestinal, dermatological, neurological, psychiatric, genitourinary, endocrinological, musculoskeletal, eye, ear, nose and throat disease, liver disorders, severe chronic kidney disease, active gastric or duodenal ulcer, benign prostate hyperplasia, phenylketonuria, hypertension, hyperthyroidism, diabetes, heart disease, aortic stenosis, tachyarrhythmia, glaucoma or phaeochromocytoma.
19. Hereditary problems of glucose-galactose malabsorption, fructose intolerance, or sucrose/isomaltase deficiency.
20. History of gastrointestinal surgery other than appendectomy.
21. Medical or surgical conditions, which might significantly interfere with the functioning of gastrointestinal tract, blood-forming organs etc.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of paracetamol, guaifenesin and phenylephrine (total) | At baseline and during 12 hours after product administration
  The maximum observed plasma concentration (Cmax)
The area under the plasma concentration-vs.-time curves from start of drug administration until the time of the last measurable concentration (AUCt) for paracetamol, guaifenesin and phenylephrine (total) | At baseline and during 12 hours after product administration
  AUCt is defined as area under the plasma concentration versus time curves from start of drug administration until the last measureable concentration.
The area under the concentration-vs.-time curve extrapolated to infinity (AUC∞) for paracetamol, guaifenesin and phenylephrine (total) | At baseline and during 12 hours after product administration
  AUC∞ is defined as area under the plasma concentration versus time curves from start of drug administration until the plasma concentration is negligible (infinity).
The extrapolated part of AUC∞, AUCExtrap of paracetamol, guaifenesin and phenylephrine (total) | From 12 hours after start of drug administration until up to 96 hours
  AUCextrap is defined as area under the plasma concentration versus time curves from 12 hours until infinity
The time at which the maximum plasma concentration is observed (tmax) for paracetamol, guaifenesin and phenylephrine (total) | At baseline and during 12 hours after product administration
  Tmax is defined as the time point at which the maximum plasma concentration (Cmax) occurs
The half-life (t1/2) for paracetamol, guaifenesin and phenylephrine (total) in plasma | At baseline and during 12 hours after product administration
  The half-life i defined as the time taken for the plasma concentration to fall to half its original value
The terminal elimination rate constant (λz) for paracetamol, guaifenesin and phenylephrine (total) in plasma | At baseline and during 12 hours after product administration
  The terminal elimination rate constant is the rate at which the drug is removed from the body system
The mean residence time (MRT) for paracetamol, guaifenesin and phenylephrine (total) | At baseline and during 12 hours after product administration
  Mean residence time (MRT) is the average amount of time that a single molecule of drug stays in the body

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of unconjugated phenylephrine | At baseline and during 12 hours after product administration
  The maximum observed plasma concentration (Cmax)
The area under the plasma concentration-vs.-time curves from start of drug administration until the time of the last measurable concentration (AUCt) for unconjugated phenylephrine | At baseline and during 12 hours after product administration
  AUCt is defined as area under the plasma concentration versus time curves from start of drug administration until the last measureable concentration.
The area under the concentration-vs.-time curve extrapolated to infinity (AUC∞) for unconjugated phenylephrine | At baseline and during 12 hours after product administration
  AUC∞ is defined as area under the plasma concentration versus time curves from start of drug administration until the plasma concentration is negligible (infinity).
The extrapolated part of AUC∞, AUCExtrap of unconjugated phenylephrine | From 12 hours after start of drug administration until up to 96 hours
  AUCextrap is defined as area under the plasma concentration versus time curves from 12 hours until the plasma concentration is negligible (infinity).
The time at which the maximum plasma concentration is observed (tmax) for unconjugated phenylephrine | At baseline and during 12 hours after product administration
  Tmax is defined as the time point at which the maximum plasma concentration (Cmax) occurs
The half-life (t1/2) for unconjugated phenylephrine in plasma | At baseline and during 12 hours after product administration
  The half-life i defined as the time taken for the plasma concentration to fall to half its original value
The terminal elimination rate constant (λz) for unconjugated phenylephrine in plasma | At baseline and during 12 hours after product administration
  The terminal elimination rate constant is the rate at which the drug is removed from the body system
The mean residence time (MRT) for unconjugated phenylephrine | At baseline and during 12 hours after product administration
  Mean residence time (MRT) is the average amount of time that a single molecule of drug stays in the body

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- Scientific Research center Eco-Safety LLC, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Redacted Study Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=12462&filename=Synopsis%20Uni_Redacted_A.pdf